CLINICAL TRIAL: NCT04278638
Title: Study of Safety and Feasibility With or Without Intraoperative Radiation in Local Advanced Laryngocarcinoma
Brief Title: IORT in Local Advanced Laryngocarcinoma
Acronym: ILAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin First Central Hospital (Other)
Responsible Party: Principal Investigator, LiLi, director of head and neck surgery division, Tianjin First Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019008
Record Dates: First submitted 2020-01-16; First posted 2020-02-20 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Laryngeal Neoplasms
MeSH Terms: conditions — Laryngeal Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with IORT (Experimental)
  Interventions: Radiation: IORT; Procedure: surgery; Radiation: External radiotherapy
- without IORT (Active Comparator)
  Interventions: Procedure: surgery; Radiation: External radiotherapy

INTERVENTIONS:
Radiation: IORT — IORT in surgery of laryngocarcinoma
  Arms: with IORT
Procedure: surgery — total laryngectomy or hemilaryngectomy
Radiation: External radiotherapy — External radiotherapy

SUMMARY:
The incidence of laryngeal cancer accounts for about 1 ~ 5% of the total body tumors. For the surgical treatment of laryngeal cancer, the development trend of laryngocarcinoma treatment is to improve the local control rate, preserve the laryngeal function of patients as far as possible, and improve the life quality of patients. The efficacy, safety and feasibility of intraoperative radiotherapy (IORT) in head and neck cancer has been demonstrated in multiple institutional (3-5) studies to optimize local control. It is still unclear whether IORT can improve the local control and have efficacy, safety and feasibility in clinic. The purpose of this study was to observe the efficacy, safety and feasibility of IORT in local advanced laryngocarcinoma .

ELIGIBILITY:
Inclusion Criteria:

1. adults over the age of 18;
2. radiographic or pathological diagnosis of local advanced laryngocarcinoma (according to NCCN guidelines);
3. the expected survival time ≥ 3 months;
4. sign informed consent for treatment and research with self-knowledge.

Exclusion Criteria:

1. there is distant metastasis;
2. pregnant women;
3. patients with CT/MRI contraindications;
4. the patient fails to receive treatment and/or follow-up as scheduled;
5. bad fluid and organ function decompensation;
6. multiple primary cancers;
7. patients participating in other trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
2-year local recurrence rate | 2 year
  In this study, no matter whether distant metastases occurred, if there was the presence of any anastomotic or lateral node recurrences, it was defined as local recurrence.
  Criteria for local recurrence include (1) MRI results suggests local tumor recurrence, (2)Laryngoscopy indicates local tumor recurrence.

SECONDARY OUTCOMES:
2-year disease free survival | 2 years
  Compare 2-year disease free survival in patients with local advanced laryngocarcinoma treated with or without IORT.
  Criteria for disease free survival means MRI and laryngoscopy (PET-CT if possible) indicate tumor free.
2-year overall survival | 2 years
  Compare 2-year overall survival in patients with local advanced laryngocarcinoma treated with or without IORT.
tissue necrosis | 2 years
  Compare the risk of tissue necrosis as determined visually by the Laryngoscope at 2 years after treatment in patients with local advanced laryngocarcinoma treated with or without IORT.
fibrosis | 2 years
  Compare the risk of fibrosis as determined visually by the Laryngoscope at 2 years after treatment in patients with local advanced laryngocarcinoma treated with or without IORT.
time of wound healing | up to 1 month
  Compare the time of wound healing after surgery in patients with local advanced laryngocarcinoma treated with or without IORT.

OTHER OUTCOMES:
pharyngeal fistula | 3 months
  Pharyngeal fistula means that saliva is stored in subcutaneous or subincisional tissues, resulting in abscess cavity rupture to the skin or incision margin, making the hypopharyngeal and esophageal lumen communicate with the skin to form a sinus tract, through which saliva or food can spill out to the skin, forming a skin fistula.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin First Central Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang Y, Li L, Zheng Y, Liu Q, Wei X, Gong X, Wang W, Lin P. A prospective, single-arm, phase II clinical trial of intraoperative radiotherapy using a low-energy X-ray source for local advanced Laryngocarcinoma (ILAL): a study protocol. BMC Cancer. 2020 Aug 6;20(1):734. doi: 10.1186/s12885-020-07233-1. PMID 32762662